CLINICAL TRIAL: NCT06237244
Title: Predicting the Presence and Severity of Coronary Artery Disease Using Surrogate Markers of Insulin Resistance: A Cross-Sectional Study
Brief Title: Insulin Resistance Indices and Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Other Study IDs: IR.SUMS.MED.REC.1402.252
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Insulin Resistance; Coronary Artery Disease
Keywords: coronary artery disease; insulin resistance; triglyceride glucose index
MeSH Terms: conditions — Insulin Resistance; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- coronary artery disease: patients with coronary angiography of at least one vessel with more than 50% stenosis
  Interventions: Diagnostic Test: triglyceride to glucose ratio; Diagnostic Test: triglycerdie to HDL ratio
- no coronary artery disease: patient with no stenosis in coronary angiography
  Interventions: Diagnostic Test: triglyceride to glucose ratio; Diagnostic Test: triglycerdie to HDL ratio

INTERVENTIONS:
Diagnostic Test: triglyceride to glucose ratio — Ratio of triglyceride level to glucose
Diagnostic Test: triglycerdie to HDL ratio — Ratio of triglyceride to HDL cholesterol

SUMMARY:
In this retrospective study from professor Kojuri clinic registry, total number of 1017 patients with first angiography were included and all data were recorded from registry. Insulin resistance was calculated using laboratory data

DETAILED DESCRIPTION:
This was an analytical cross-sectional retrospective study involving patients with suspected CAD who underwent coronary angiography between December 2018 and May 2023. The information was obtained from patients referred to the outpatient cardiovascular clinic (Professor Kojuri Cardiology Clinic, Shiraz, Iran, www.kojuriclinic.com). Data was extracted from Professor Kojuri Cardiology Clinic database, including patient's information about the clinical history, presence or absence of specific diseases, angiography/angioplasty results, medications, and laboratory values.

A total of 14,708 patients who had undergone coronary angiography at least once were examined. After applying exclusion criteria, 1017 eligible cases were selected for data analysis.

The following data was recorded for the included patients: demographic data, past medical history (such as DM, hypertension, etc.), systolic and diastolic blood pressure, weight and height, fasting plasma glucose (FPG), hemoglobin A1c (HbA1c), total cholesterol (TC), triglyceride (TG), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), and serum creatinine (Cr). Body mass index (BMI) was calculated as weight (Kg) divided by the square of height (m2). Obesity was defined as BMI ≥ 30 Kg/m2.

Laboratory values were selected from the time before angiography, and if not available, from the time shortly after the angiography. This helped us find those values which could best represent the metabolic state of patients at the time of angiography, while reducing the confounding effect of statin use.

ELIGIBILITY:
Inclusion Criteria:

* patients with age more than 18 years and having undergone coronary angiography

Exclusion Criteria:

* incomplete data
* history of prior coronary angiography or revascularization (percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG))
* serum creatinine > 1.4 mg/dL
* history of chronic kidney disease (CKD)
* cancer,

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients more than 18 years old referred for evaluation of coronary artery disease for their first time
Sampling Method: Non-Probability Sample
Enrollment: 1017 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
insulin resistance index: level of triglyceride to glucose ratio from blood sample | 3 years
  correlation of coronary artery disease and triglyceride glucose ratio in blood laboratory tests
insulin resistance index: Level of triglyceride to HDL ratio from blood sample | 3 years
  correlation of coronary artery disease and triglyceride to HDL level ratio in blood laboratory sample

SECONDARY OUTCOMES:
metabolic syndrome | 3 years
  metabolic syndrome based on criteria of metabolic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Javad Kojuri, MD. MS., Principal Investigator — Professor kojuri cardiology clinic
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: No
Data are available based on rational request

REFERENCES:
- [Derived] Jahangiri S, Mosalamiaghili SA, Heydarzadeh R, Yousefzadeh M, Golchin Vafa R, Zarifkar H, Assadian K, Sohrabizadeh S, Zarifkar H, Sadeghi M, Hosseini N, Montaseri M, Hosseini SA, Kojuri J. Predicting the presence and severity of coronary artery disease using surrogate markers of insulin resistance: A cross-sectional study. ARYA Atheroscler. 2025;21(1):44-53. doi: 10.48305/arya.2025.42573.2960. PMID 40401209